CLINICAL TRIAL: NCT01034189
Title: A Phase II Study of Combining Cetuximab Plus Twice Weekly Paclitaxel/Cisplatin Concurrent Chemoradiotherapy (TP-CCRT) Followed With or Without Esophagectomy for Loco-regional Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Cetuximab/Paclitaxel/Cisplatin Concurrent Chemoradiotherapy Followed by Esophagectomy for Loco-regional Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chih-Hung Hsu / Department of Oncology, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200803088M
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Chemoradiotherapy; Paclitaxel; Cetuximab
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cetuximab; Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targeted therapy (Experimental): Concurrent chemoradiotherapy with cetuximab, paclitaxel, and cisplatin followed by, if feasible, esophagectomy
  Interventions: Drug: Cetuximab; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cetuximab — Cetuximab: loading dose 400 mg/m2, 2h- IVF, 3~ 5 days prior to starting CCRT (on week-1); followed by 250 mg/m2/ week, 1h- IVF, for 4 weeks (i.e., week 1 to week 4. during CCRT).
  Other Names: Erbitux
Drug: Paclitaxel — T: Paclitaxel 35 mg/m2, 1h IVF, on day 1 and day 4 of each week, week1 to week4 during CCRT.
Drug: Cisplatin — P: Cisplatin 15 mg/m2, 1 h IVF, on day 2 and day 5 of each week, week1 to week4 during CCRT.
Radiation: Radiotherapy — Radiotherapy: (three-dimensional conformal radiotherapy or intensity modulated radiotherapy) 200 cGy/fraction, once daily, 5 days a week, to a total dose of 4000 cGy.

SUMMARY:
We hypothesize that the addition of cetuximab to twice weekly paclitaxel/cisplatin concurrent chemoradiotherapy (TP-CCRT) as the adjunctive therapy before esophagectomy or as a definitive CRT would improve the therapeutic efficacy of TP-CCRT in patients with loco-regional esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
We hypothesize that the addition of cetuximab to twice weekly paclitaxel/cisplatin concurrent chemoradiotherapy as the adjunctive therapy before esophagectomy or as a definitive CRT would improve the therapeutic efficacy of TP-CCRT in patients with loco-regional esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven squamous cell carcinoma of esophagus.
2. Loco-regional diseases, which are defined by TNM system of American Joint Committee on Cancer (AJCC) Cancer Staging System (6th edition) in 2002, fulfilling one of the following criteria:

   A. T3, N0, M0; B. T1-3, N1, M0; C. T1-3 or N0-1, M1a will be eligible provided the lesions could be covered by appropriate radiation fields.
3. Age ≥ 18 years old.
4. Performance status ECOG 0~2.
5. Adequate bone marrow reserves, defined as:

   A. white blood cells (WBC) ≥ 4,000/µl or neutrophil count (ANC) ≥ 2,000/µl; B. platelets ≥ 100,000/µl.
6. Adequate liver function reserves, defined as:

   A. hepatic transaminases ≤ 2.5 x upper limit of normal (ULN); B. serum total bilirubin ≤ 1.5 x upper limit of normal (ULN).
7. Adequate renal function: Creatinine ≤1.5 mg/dl
8. Written informed consent.

Exclusion Criteria:

1. Invasion to surrounding organ (T4 disease).
2. Distant metastasis, except M1a disease listed in the inclusion criteria 2-C.
3. Adenocarcinoma of gastroesophageal (GE) junction.
4. Prior thoracic irradiation.
5. Synchronously diagnosed squamous cell carcinoma of aerodigestive way, other than esophageal cancer.
6. Prior malignancy, except for the following:

   A. adequately treated basal cell or squamous cell skin cancer; B. in-situ cervical cancer; C. Note: previously treated aerodigestive squamous cell carcinoma is not allowed.
7. Significant co-morbid disease, which prohibit the conduction of chemotherapy, concurrent chemoradiotherapy, or radical surgery, such as active systemic infection, symptomatic cardiac or pulmonary disease, or psychiatric disorders.
8. Estimated life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
To determine the clinical response rate in patients with loco-regional esophageal squamous cell carcinoma treated with cetuximab combined with twice weekly paclitaxel/cisplatin concurrent chemoradiotherapy (C-TP-CCRT, 40 Gy). | 2 years

SECONDARY OUTCOMES:
Pathologic complete response (pCR). | 2 years
Disease-free survival. | 2 years
Safety and toxicity of cetuximab combined with twice weekly TP-CCRT, followed by surgery. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Chie Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Guo JC, Huang TC, Lin CC, Hsieh MS, Chang CH, Huang PM, Lee JM, Hsu FM, Chia-Hsien Cheng J, Wang HP, Yeh KH, Cheng AL, Hsu CH. Postchemoradiotherapy Pathologic Stage Classified by the American Joint Committee on the Cancer Staging System Predicts Prognosis of Patients with Locally Advanced Esophageal Squamous Cell Carcinoma. J Thorac Oncol. 2015 Oct;10(10):1481-9. doi: 10.1097/JTO.0000000000000651. PMID 26313683